CLINICAL TRIAL: NCT02757131
Title: Dedicated Ambulator-assisted Physical Activity to Improve Hospital Outcome Measures in Elderly Patients: A Randomized, Controlled Trial
Brief Title: Dedicated Ambulator-assisted Physical Activity to Improve Hospital Outcome Measures in Elderly Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Aaron Hamilton, Staff Physician, The Cleveland Clinic
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-335
Record Dates: First submitted 2016-04-19; First posted 2016-04-29 (Estimated); Last update posted 2017-08-10 (Actual); Status verified 2017-08

CONDITIONS: Weakness; Hospital Acquired Condition
Keywords: Mobility; Elderly; Hospitalized patient
MeSH Terms: conditions — Asthenia; Iatrogenic Disease | interventions — Walking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Patients randomized to the intervention group will be asked to participate in the ambulation protocol outlined by the Physical Therapy (PT) staff 3 times daily under the supervision of the dedicated ambulator PCNA.
  The ambulator will be trained by the physical therapy team on how to implement the protocol prior to initiation of the study.
  Interventions: Other: Ambulation
- Control (No Intervention): The cohort of patients randomized to "usual care" will not be seen by the dedicated ambulator, but will not otherwise be restricted in nursing's baseline ability to execute nursing specific recommendations placed by the PT team.

INTERVENTIONS:
Other: Ambulation — Patients randomized to the intervention group will be asked to participate in the ambulation protocol outlined by the PT staff 3 times daily under the supervision of the dedicated ambulator PCNA. This protocol will involve four exercise levels (mobilization, standing, walking, stairs) that may be implemented depending on the current physical capacity of the patient. The cohort of patients randomized to "ambulator protocol" will also receive the usual care by primary nursing.
  In an effort to best characterize mobility in these patients, the team will collect Braden Scale Activity data from the electronic health record, and provide each patient a mobility tracking device to directly record daily steps taken while the patient is in the hospital. Daily step counts will be collected on a weekly basis from each device. The Braden Scale is entered by nursing on each patient at least daily and measures current activity level on a 4-point scale.
  Arms: Intervention

SUMMARY:
Bedrest and lack of mobility in the inpatient hospital setting hastens the functional decline of elderly patients and is associated with increased risk of complications such as falls, delirium, venous thrombosis, and skin breakdown. These adverse health effects drive increased cost as patients spend additional time in both the acute (hospital) and post-acute care settings. Physical activity is thus widely recognized as an important factor for improving outcomes in hospitalized patients; however, numerous challenges to its implementation exist. Specifically, although it has been found that with small increases in physical activity such as increasing number of steps by only 600 daily for inpatients, length of stay can be reduced by nearly 2 days, usual care in many hospitals, including the Cleveland Clinic, does not include exercise, and physicians do not all regularly order physical activity for their hospitalized patients. Even when activity is recommended or ordered, compliance and execution of the orders has been spotty and/or negligible. It is therefore clear that the current system for the provision of ambulation is ineffective. The investigators hypothesize that a graded protocol of ambulation which can be implemented by a dedicated patient care nursing assistant (PCNA) multiple times daily will provide significant benefit to patients without the labor and cost requirements of full-time nursing and physical therapy expertise. The objective of this study is to assess the feasibility and effectiveness of dedicated ambulator-assisted physical activity in elderly inpatients. The primary hypothesis is that an ambulator-assisted intervention for hospitalized elderly inpatients will prove feasible and may result in improved hospital outcomes, including less need for inpatient rehabilitation and shorter length of stay in the hospital. This study will provide pilot data for a larger randomized trial.

DETAILED DESCRIPTION:
Specific Aims

Aim 1: To determine the feasibility of implementing an ambulator-assisted exercise intervention in elderly patients on an inpatient medicine service.

The investigators will work closely with the physical therapy team to develop a graded ambulation protocol that can be implemented multiple times daily per enrolled patient by a PCNA. Investigators will work closely with the medicine units to recruit eligible patients and assess protocol implementation including recruitment, patient cooperation, and scheduling.

Aim 2: To determine the effects of an ambulator-assisted exercise intervention on discharge disposition, length of stay and cost.

The investigators will measure the proportion of patients in the intervention and usual care group who are discharged to home vs. acute rehabilitation facilities. Length of stay and cost will be obtained from hospital billing records.

Research Strategy

The investigators propose the development of a feasible program to assist in improving the physical capacity of elderly inpatients. Such improvements may translate to cost savings in the form of decreased length of stay, improved discharge disposition, and fewer hospital-related complications, but establishing that is not the purpose of this study. The investigators propose that the most feasible and cost-effective implementation of such a program will utilize a patient care nursing assistant (PCNA) dedicated to carrying out a graded ambulation protocol in eligible patients multiple times daily. A simple and standardized protocol for ambulation will reduce the need for the expertise of a dedicated physical therapist. Additionally, utilizing an existing mechanism for assessing baseline functional capacity, the 6-Clicks score, will eliminate the time and personnel requirements for evaluation of patient eligibility. This score has been validated as a mechanism to assess patient mobility limitations in an acute care setting and is currently used on all patients seen by physical therapy on the inpatient medicine services.

This pilot study will enable the investigators to identify which patients would tolerate the intervention and what degree of participation would be meaningful to improve the outcomes measured. The study will begin by enrolling patients with 6-Clicks scores of 16-20, as these patients will experience the greatest benefit from an ambulation protocol. At present, such patients do not receive any PT intervention and ambulation by nurses occurs only sporadically as time allows. Additionally, the pilot will help to bring clarity to the direct impact of aggressive mobilization of medical inpatients on important outcomes that are directly tied to healthcare cost. Results of this work will inform feasibility and power calculations for a larger randomized trial. Results of that trial could directly impact the approach to the medical inpatient in terms of prioritizing and resourcing mobilization strategies.

Preliminary findings from this pilot study demonstrating the feasibility of a dedicated ambulator-assisted physical activity protocol and its potential impact on hospital outcomes will provide the justification for external funding of a larger randomized clinical trial. Lessons learned from the pilot study will allow us to optimize the ambulation protocol and target population for a larger study. Such a study would investigate the effect of the ambulator-assisted physical activity protocol on patient mobility associated health care costs. This work could shift the current paradigm that aggressive mobilization is reserved for post-acute care settings and could serve as a model for improving the value of care provided to elderly patients in acute care facilities.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women 60 years of age or older admitted as inpatients to floors G80, H80, H81 and G81 in the Medicine Institute, Cleveland Clinic Main Campus during the study time period
2. Hospitalized for a medical illness
3. Complete history and physical examination on file
4. Physical therapy consult and 6-Clicks score between 16-20 a. This is based on a usual care assessment ordered by a physician that will happen prior to any study recruitment - it is entirely independent of the study

Exclusion Criteria:

1. Observational status
2. Admission to ICU
3. Surgical patients
4. Patients diagnosed with: decompensated heart failure, unstable angina, other medical conditions precluding participation in exercise/ambulation
5. Comfort care measures only

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Discharge disposition from hospitalization - from electronic health record | Will be measured at time of discharge for each patient through study completion, up to six weeks
  The investigators will track the care setting patients are discharged to from the inpatient stay. This will include home, home with home health care, skilled nursing facility, acute rehab, nursing home, hospice
Length of stay in days for participant's hospitalization | Will be measured at the time of discharge for each patient through study completion, up to six weeks
  Time, in days, elapsed from patient admission to discharge

SECONDARY OUTCOMES:
Patient in-hospital mortality | Will be measured for the episode of care associated with the admission the patient was enrolled in the study, up to six weeks
Admission to Intensive care unit after initiation of intervention - from electronic health record | Will be measured at patient level at the completion of each patient discharge, up to six weeks
  Participants enrolled in the study will be followed and if their care is escalated to an intensive care unit, the investigators will track
Participant inpatient falls - binary yes/no extracted from the safety event reporting system which closely tracks all inpatient falls | Will be measured at the time of discharge for the patient and will include any fall during the index admission
New onset of stroke, Deep Vein Thrombosis, Pulmonary embolus or pneumonia during hospitalization as determined by billing codes for participants | Will be measured at patient level for each admission and will end at discharge, up to six weeks
  Participants with billing codes for the above conditions that are not present on admission will be included in the outcome measure.
Readmission within 30 days | 30 days after discharge
Change in 6-Clicks score from admission to discharge - as measured by the physical therapy team with each visit - this is extracted from our electronic health record | Will be measured at patient level for each admission and will end at discharge, up to six weeks
  The 6-clicks score is a validated marker of mobility for inpatients

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Hamilton, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Foundation, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] National Center for Health Statistics (US). Health, United States, 2013: With Special Feature on Prescription Drugs. Hyattsville (MD): National Center for Health Statistics (US); 2014 May. Report No.: 2014-1232. Available from http://www.ncbi.nlm.nih.gov/books/NBK209224/ PMID 24967476
- [Background] Corcoran PJ. Use it or lose it--the hazards of bed rest and inactivity. West J Med. 1991 May;154(5):536-8. PMID 1866946
- [Background] Zisberg A, Shadmi E, Sinoff G, Gur-Yaish N, Srulovici E, Admi H. Low mobility during hospitalization and functional decline in older adults. J Am Geriatr Soc. 2011 Feb;59(2):266-73. doi: 10.1111/j.1532-5415.2010.03276.x. PMID 21314647
- [Background] Gillick MR, Serrell NA, Gillick LS. Adverse consequences of hospitalization in the elderly. Soc Sci Med. 1982;16(10):1033-8. doi: 10.1016/0277-9536(82)90175-7. PMID 6955965
- [Background] Hirsch CH, Sommers L, Olsen A, Mullen L, Winograd CH. The natural history of functional morbidity in hospitalized older patients. J Am Geriatr Soc. 1990 Dec;38(12):1296-303. doi: 10.1111/j.1532-5415.1990.tb03451.x. PMID 2123911
- [Background] Sager MA, Franke T, Inouye SK, Landefeld CS, Morgan TM, Rudberg MA, Sebens H, Winograd CH. Functional outcomes of acute medical illness and hospitalization in older persons. Arch Intern Med. 1996 Mar 25;156(6):645-52. PMID 8629876
- [Background] Heit JA, Silverstein MD, Mohr DN, Petterson TM, O'Fallon WM, Melton LJ 3rd. Risk factors for deep vein thrombosis and pulmonary embolism: a population-based case-control study. Arch Intern Med. 2000 Mar 27;160(6):809-15. doi: 10.1001/archinte.160.6.809. PMID 10737280
- [Background] Campbell AJ, Borrie MJ, Spears GF. Risk factors for falls in a community-based prospective study of people 70 years and older. J Gerontol. 1989 Jul;44(4):M112-7. doi: 10.1093/geronj/44.4.m112. PMID 2738307
- [Background] Fisher SR, Kuo YF, Graham JE, Ottenbacher KJ, Ostir GV. Early ambulation and length of stay in older adults hospitalized for acute illness. Arch Intern Med. 2010 Nov 22;170(21):1942-3. doi: 10.1001/archinternmed.2010.422. No abstract available. PMID 21098357
- [Background] Graf C. Functional decline in hospitalized older adults. Am J Nurs. 2006 Jan;106(1):58-67, quiz 67-8. doi: 10.1097/00000446-200601000-00032. PMID 16481783
- [Background] Chang JT, Morton SC, Rubenstein LZ, Mojica WA, Maglione M, Suttorp MJ, Roth EA, Shekelle PG. Interventions for the prevention of falls in older adults: systematic review and meta-analysis of randomised clinical trials. BMJ. 2004 Mar 20;328(7441):680. doi: 10.1136/bmj.328.7441.680. PMID 15031239
- [Background] Lazarus BA, Murphy JB, Coletta EM, McQuade WH, Culpepper L. The provision of physical activity to hospitalized elderly patients. Arch Intern Med. 1991 Dec;151(12):2452-6. PMID 1747003
- [Background] McVey LJ, Becker PM, Saltz CC, Feussner JR, Cohen HJ. Effect of a geriatric consultation team on functional status of elderly hospitalized patients. A randomized, controlled clinical trial. Ann Intern Med. 1989 Jan 1;110(1):79-84. doi: 10.7326/0003-4819-110-1-79. PMID 2642284
- [Background] Said CM, Morris ME, Woodward M, Churilov L, Bernhardt J. Enhancing physical activity in older adults receiving hospital based rehabilitation: a phase II feasibility study. BMC Geriatr. 2012 Jun 8;12:26. doi: 10.1186/1471-2318-12-26. PMID 22676723
- [Background] Inouye SK, Wagner DR, Acampora D, Horwitz RI, Cooney LM Jr, Tinetii ME. A controlled trial of a nursing-centered intervention in hospitalized elderly medical patients: the Yale Geriatric Care Program. J Am Geriatr Soc. 1993 Dec;41(12):1353-60. doi: 10.1111/j.1532-5415.1993.tb06487.x. PMID 8227919
- [Background] Timmerman RA. A mobility protocol for critically ill adults. Dimens Crit Care Nurs. 2007 Sep-Oct;26(5):175-9; quiz 180-1. doi: 10.1097/01.DCC.0000286816.40570.da. PMID 17704667
- [Background] Morris PE, Goad A, Thompson C, Taylor K, Harry B, Passmore L, Ross A, Anderson L, Baker S, Sanchez M, Penley L, Howard A, Dixon L, Leach S, Small R, Hite RD, Haponik E. Early intensive care unit mobility therapy in the treatment of acute respiratory failure. Crit Care Med. 2008 Aug;36(8):2238-43. doi: 10.1097/CCM.0b013e318180b90e. PMID 18596631
- [Background] Jette DU, Stilphen M, Ranganathan VK, Passek SD, Frost FS, Jette AM. Validity of the AM-PAC "6-Clicks" inpatient daily activity and basic mobility short forms. Phys Ther. 2014 Mar;94(3):379-91. doi: 10.2522/ptj.20130199. Epub 2013 Nov 14. PMID 24231229